CLINICAL TRIAL: NCT04100317
Title: Result of Spanning Bridge Plate Fixation for Comminuted Intra Articular Distal Radial Fractures.
Brief Title: Spanning Bridged Plate in Comminuted Distal Radius Fractures
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Anass Abdeslam kabbour Hanzaz, Dr, Assiut University
Other Study IDs: Bpf in distal radius fractures
Record Dates: First submitted 2019-09-20; First posted 2019-09-24 (Actual); Last update posted 2019-09-24 (Actual); Status verified 2019-09

CONDITIONS: Distal Radius Fracture
Keywords: Pridge plate
MeSH Terms: conditions — Wrist Fractures

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This study To evaluate the result of using spanning bridge plate in comminuted distal radius fractures.

DETAILED DESCRIPTION:
Distal radius fractures are the most common long bone fracture and the incidence appears to be increasing worldwide. They have been found to account for approximately 17% of all fracture-related emergency department visits. These types of injuries have a bimodal age distribution. The first peak represents young patients involved in high energy traumas, and the second peak represents elderly patients with lower to moderate energy injuries secondary to osteoporosis.Surgical treatment for distal radius fractures varies, as there are numerous techniques for fixation. The goals of fixation are anatomic reduction and stability, as this has been shown to result in improved chances for functional recovery . The use of volar locking plateshas become the standard for treatment of the majority of distal radius fractures requiring surgery . However, adequate fixation for high energy comminuted fractures with or without metadia-physeal extension remains a major treatment challenge. Severely comminuted articular fractures are technically challenging in terms of obtaining an adequate reduction and achieving stabilization with a standard periarticular volar plating technique. The small fracture fragments are often not able to be stabilized with the screws from the volar plate, and the proximally-oriented tension from the forearm musculature acts to pull on the carpus causing further collapse of the articular surface. As an alternate to the volar plate, these types of injuries have been historically treated with an external fixator with or without Kirschner wires. However, it has been reported that highly comminuted distal radius fractures are associated with a 52%-63% complication rate when treated with external fixation . Therefore, despite poor fixation capabilities withthese fracturetypes,thevolarplate remainsthego-to devicefor most surgeons when faced with comminuted articular distal radial fractures. In these circumstances, the dorsal distraction plate (also called dorsal "bridge" plating technique) can serve as an improved fixation technique by allowing comminuted articular fragments to reduce under ligamentotaxis and provide a buttress for the dorsal cortex of the distal radius. In addition, a long dorsal plate can bridge past metaphyseal comminution, which cannot be so easily addressed with standard volar plating . The bridge plate can also be left in place for an extended period of time without the risk of the aforementioned complications of prolonged external fixation use . Finally, the dorsal distraction plate is technically a much easier operation to perform than volar plating for complex articular fractures. Recently, there has been increased use of dorsal distraction plating for these types of injuries .

ELIGIBILITY:
Inclusion Criteria:

* age 18-60 years old
* early trouma (within two weeks)

Exclusion Criteria:

* open fractures
* concomitant limb injuries
* old fractures more than two weeks
* sever osteoporosis and osteopenia.

Ages: 18 Years to 60 Years | Sex: All
Age Groups: Adult
Study Population: Troumatized population with age 18 to 60 years old with comminuted intra articular distal radius fractures.
Sampling Method: Non-Probability Sample
Enrollment: 20 (Estimated)
Dates: Start 2019-09-20 (Estimated); Primary Completion 2020-09-20 (Estimated); Study Completion 2020-10-20 (Estimated)

PRIMARY OUTCOMES:
Wrist range of movement | Baseline
  Degree measurment of wrist Flexion. Extension radial and ulnur deviatin

SECONDARY OUTCOMES:
Radilogical parameters | Baseline
  By taking new xrays and exactly calculate the distal radius angels and parameters by calculate the exact deviatin
Grip strength | Baseline
  By using grip strength power
Union | Baseline
  Assesment of union condition by Dexa scan

CONTACTS AND LOCATIONS:
Overall Officials: Amr Pr Elsayed, Study Director — Proffissor

REFERENCES:
- [Background] Matullo KS, Dennison DG. Outcome following distally locked volar plating for distal radius fractures with metadiaphyseal involvement. Hand (N Y). 2015 Jun;10(2):292-6. doi: 10.1007/s11552-014-9713-z. PMID 26034446
- [Background] Geller L, Bernstein M, Carli A, Berry G, Reindl R, Harvey E. Efficacy of different fixation devices in maintaining an initial reduction for surgically managed distal radius fractures. Can J Surg. 2009 Oct;52(5):E161-6. PMID 19865547
- [Background] Mann T, Lee DJ, Dahl J, Elfar JC. Can Radiocarpal-Spanning Fixation Be Made More Functional by Placing the Wrist in Extension? A Biomechanical Study Under Physiologic Loads. Geriatr Orthop Surg Rehabil. 2016 Mar;7(1):23-9. doi: 10.1177/2151458515621109. PMID 26929853